CLINICAL TRIAL: NCT00824382
Title: Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 4 Weeks of Once Daily Treatment of Orally Inhaled BI 1744 CL Delivered by the Respimat Inhaler in Japanese Patients With COPD
Brief Title: Efficacy and Safety of 4 Weeks Treatment With Inhaled BI 1744 CL in Japanese Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.22
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (4):
- BI 1744 CL 5 Âµg (Experimental): 2 puffs of 2.5 Âµg/actuation
  Interventions: Drug: BI 1744 CL 5 Âµg
- BI 1744 CL 10 Âµg (Experimental): 2 puffs of 5 Âµg/actuation
  Interventions: Drug: BI 1744 CL 10 Âµg
- Placebo (Placebo Comparator): 2 puffs
  Interventions: Drug: Placebo
- BI 1744 CL 2 Âµg (Experimental): 2 puffs of 1 Âµg/actuation
  Interventions: Drug: BI 1744 CL 2 Âµg

INTERVENTIONS:
Drug: BI 1744 CL 2 Âµg — 2 puffs of 1 Âµg/actuation delivered by the RespimatÂ® inhaler
  Arms: BI 1744 CL 2 Âµg
Drug: BI 1744 CL 5 Âµg — 2 puffs of 2.5 Âµg/actuation delivered by the RespimatÂ® inhaler
  Arms: BI 1744 CL 5 Âµg
Drug: BI 1744 CL 10 Âµg — 2 puffs of 5 Âµg/actuation delivered by RespimatÂ®
  Arms: BI 1744 CL 10 Âµg
Drug: Placebo — 2 puffs delivered by the RespimatÂ® inhaler
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the optimum dose(s) of BI 1744 CL inhalation solution delivered by the Respimat inhaler once daily for 4 weeks in Japanese patients with chronic obstructive pulmonary disease (COPD). The selection of the optimum dose(s) will be based on bronchodilator efficacy, safety evaluations and pharmacokinetic evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with GCP guidelines prior to participation in the trial.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria: Patients must have relatively stable, moderate to severe airway obstruction with a post-bronchodilator FEV1 >=30% of predicted normal and <80% of predicted normal and a post-bronchodilator FEV1/FVC <70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years. Pack-Years = [Number of cigarettes/day/20] - years of smoking Patients who have never smoked cigarettes must be excluded.
5. Patients must be able to perform technically acceptable pulmonary function tests (both supervised and unsupervised) and PEFR measurements, and must be able to record a patient diary during the study period as required in the protocol.
6. Patients must be able to inhale medication in a competent manner from the Respimat inhaler and from a MDI.

Exclusion Criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may i) put the patient at risk because of participation in the study ii) influence the results of the study, or iii) cause concern regarding the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an AST >80 IU/L, ALT >80 IU/L, bilirubin >1.5 x ULN or creatinine >1.5 x ULN will be excluded regardless of clinical condition (a repeat laboratory evaluation will not be conducted in these patients)
3. Patients with a history of asthma or a total blood eosinophil count >=600/mm3. A repeat eosinophil count will not be conducted in these patients
4. Patients with any of the following conditions:

   * a diagnosis of thyrotoxicosis
   * a diagnosis of paroxysmal tachycardia (>100 beats per minute)
   * a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms) as recommended by ICH E14. For patients who have a QTc interval between 450 ms and 500 ms, as judged by site personnel, there will be a confirmatory reading by centralized evaluation institute. If the confirmatory reading is still greater than 450 ms, patient will be excluded. Patients with a QTc interval >=500 ms will immediately be excluded from the study.
   * a history of additional risk factors for Torsade de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT Syndrome) as recommended by ICH E14.
5. Patients with any of the following conditions:

   * a history of myocardial infarction within 1 year
   * a diagnosis of clinically relevant cardiac arrhythmia
   * known active tuberculosis
   * a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last 5 years (patients with treated basal cell carcinoma are allowed)
   * a history of life-threatening pulmonary obstruction
   * a history of cystic fibrosis
   * clinically evident bronchiectasis
   * a history of significant alcohol or drug abuse
6. Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1)
7. Patients being treated with any of the following concomitant medications:

   * medications that prolong the QT/QTc interval
   * oral beta-adrenergics and beta-adrenergics patchs
   * beta-blockers (topical beta-blockers for ocular conditions are allowed)
   * oral corticosteroid medication at unstable doses (i.e. less than 6 weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
8. Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
9. Patients who have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
10. Patients who have taken an investigational drug within 1 month or 6 half lives (whichever is greater) prior to screening visit
11. Patients with known hypersensitivity to beta-adrenergics drugs, BAC, EDTA or any other component of the Respimat inhalation solution delivery system
12. Pregnant or suspect of pregnant or women who are willing to become pregnant during the study period or nursing women
13. Patients who have previously been participated in this study or are currently participating in another study
14. Patients who are unable to comply with pulmonary medication restrictions prior to randomisation
15. The randomization of patients with any respiratory infection or COPD exacerbation in the 6 weeks prior to the screening visit or during the screening period should be postponed. Patients may be randomised 6 weeks following recovery from the infection or exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (48):
- Japan (48):
  - 1222.22.048 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 1222.22.044 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 1222.22.008 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1222.22.002 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1222.22.041 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1222.22.027 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1222.22.028 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1222.22.018 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1222.22.021 Boehringer Ingelheim Investigational Site, Hitachi, Ibaraki
  - 1222.22.010 Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaraki
  - 1222.22.012 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1222.22.009 Boehringer Ingelheim Investigational Site, Kamogawa, Chiba
  - 1222.22.023 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1222.22.025 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1222.22.017 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 1222.22.004 Boehringer Ingelheim Investigational Site, Kitakyusyu, Fukuoka
  - 1222.22.020 Boehringer Ingelheim Investigational Site, Koga, Fukuoka
  - 1222.22.014 Boehringer Ingelheim Investigational Site, Komaki, Aichi
  - 1222.22.032 Boehringer Ingelheim Investigational Site, Kumamoto, Kumamoto
  - 1222.22.005 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1222.22.029 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1222.22.033 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1222.22.050 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1222.22.022 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1222.22.015 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1222.22.043 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1222.22.001 Boehringer Ingelheim Investigational Site, Naka-gun, Ibaraki
  - 1222.22.007 Boehringer Ingelheim Investigational Site, Niigata, Niigata
  - 1222.22.040 Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - 1222.22.042 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1222.22.034 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1222.22.038 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1222.22.049 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1222.22.045 Boehringer Ingelheim Investigational Site, Osaka-sayama, Osaka
  - 1222.22.019 Boehringer Ingelheim Investigational Site, Sakai, Oasaka
  - 1222.22.006 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1222.22.051 Boehringer Ingelheim Investigational Site, Sashima-gun, Ibaraki
  - 1222.22.031 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1222.22.013 Boehringer Ingelheim Investigational Site, Seto, Aichi
  - 1222.22.024 Boehringer Ingelheim Investigational Site, Shibata-gun, Miyagi
  - 1222.22.003 Boehringer Ingelheim Investigational Site, Takarazuka, Hyogo
  - 1222.22.026 Boehringer Ingelheim Investigational Site, Tsukuba, Ibaraki
  - 1222.22.030 Boehringer Ingelheim Investigational Site, Ube, Yamaguchi
  - 1222.22.037 Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - 1222.22.047 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - 1222.22.016 Boehringer Ingelheim Investigational Site, Yamagata, Yamagata
  - 1222.22.036 Boehringer Ingelheim Investigational Site, Yao, Osaka
  - 1222.22.011 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Derived] Ichinose M, Takizawa A, Izumoto T, Tadayasu Y, Hamilton AL, Kunz C, Fukuchi Y. Efficacy and safety of the long-acting beta2-agonist olodaterol over 4 weeks in Japanese patients with chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2015 Aug 20;10:1673-83. doi: 10.2147/COPD.S86002. eCollection 2015. PMID 26316741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled in the trial on 13 January 2009 and the last patient made the last visit on 31 March 2010. A total of 515 patients were enrolled in the trial at 48 trial sites. Of the 515 patients, 328 patients were entered in the trial and were randomly assigned to receive either one of the four treatments for 4 weeks.
Pre-assignment Details: Informed consent was obtained prior to patient participation in the trial, which included medication washout procedures or restrictions. Upon obtaining consent, the patients were instructed on the medication washout and other restrictions for the screening PFT (Visit 1).
Groups:
- Placebo: Placebo
- Olodaterol 2mcg: Olodaterol 2mcg inhalation solution via Respimat
- Olodaterol 5mcg: Olodaterol 5mcg inhalation solution via Respimat
- Olodaterol 10mcg: Olodaterol 10mcg inhalation solution via Respimat
Period: Overall Study
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Started | 79 | 84 | 79 | 86
Completed | 74 | 82 | 76 | 81
Not Completed | 5 | 2 | 3 | 5
Not completed — Adverse Event | 4 | 1 | 1 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Investigator's decision | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The treated set consisting of all randomised patients for whitch at least one investigational treatment was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg | Total
Number analyzed (Participants) | 79 | 84 | 79 | 86 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.5) | 68.9 (7.6) | 70.1 (6.7) | 69.3 (7.4) | 69.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 6 | 18
  Male | 75 | 79 | 76 | 80 | 310
Percent predicted normal FEV1 [Mean (Standard Deviation); unit: percent] — Based on Japanese equation
  percent | 50.64 (12.32) | 51.36 (14.15) | 52.07 (12.82) | 51.73 (11.81) | 51.45 (12.76)
Percent predicted normal FEV1 [Number; unit: Participants] — based on Japanese equation
  Participants
    < 30% | 1 | 1 | 0 | 0 | 2
    30 to < 50% | 35 | 40 | 38 | 41 | 154
    50% to 80% | 43 | 43 | 41 | 45 | 172

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 Response at Week 4
Description: The change from baseline in trough FEV1 after 4 weeks of treatment. Trough FEV1 is defined as the mean of the two FEV1 values (performed at -1 hour and -10 minutes prior to next test-drug inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FEV1 response is defined as the change from baseline . Baseline trough FEV1 is the mean of the two pre-treatment FEV1 values measured at Visit 2 prior to administration of the first dose of study medication.
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | -0.032 (0.015) | 0.059 (0.015) | 0.100 (0.015) | 0.100 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.091, 95% CI [0.051 to 0.131], Standard Error of Mean 0.020
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.132, 95% CI [0.091 to 0.172], Standard Error of Mean 0.021
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.132, 95% CI [0.092 to 0.172], Standard Error of Mean 0.020

2. Secondary Outcome: Trough FEV1 Response at Week 2
Description: Trough FEV1 is defined as the mean of the two FEV1 values (performed at -1 hour and -10 minutes prior to next test-drug inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FEV1 response is defined as the change from baseline in trough FEV1. Baseline trough FEV1 is the mean of the two pre-treatment FEV1 values measured at Visit 2 prior to administration of the first dose of study medication
Time Frame: baseline and after 2 weeks treatment
Population: The full analysis set (FAS) - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | -0.020 (0.016) | 0.061 (0.015) | 0.120 (0.016) | 0.136 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p = 0.0002, ANCOVA; Based on an analysis of covariance with terms for baseline, treatment and center (center random, all other effects fixed); Mean Difference (Final Values) = 0.081, 95% CI [0.039 to 0.124], Standard Error of Mean 0.021 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.098 to 0.184], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.157, 95% CI [0.115 to 0.199], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo

3. Secondary Outcome: FEV1 AUC(0-3) Response at 4 Weeks
Description: The change from baseline in FEV1 AUC(0-3) after 4 weeks of treatment. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in liters.
  Due to normalization the unit is liters.
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | -0.020 (0.017) | 0.118 (0.016) | 0.177 (0.017) | 0.173 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.138, 95% CI [0.095 to 0.182], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.197, 95% CI [0.154 to 0.241], Standard Error of Mean 0.022
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.193, 95% CI [0.150 to 0.236], Standard Error of Mean 0.022

4. Secondary Outcome: FEV1 Peak(0-3) Response at 4 Weeks
Description: The change from baseline in FEV1 peak(0-3) after 4 weeks of treatment.
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | 0.025 (0.017) | 0.170 (0.017) | 0.227 (0.017) | 0.220 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.146, 95% CI [0.101 to 0.191], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.202, 95% CI [0.157 to 0.247], Standard Error of Mean 0.023
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.196, 95% CI [0.151 to 0.240], Standard Error of Mean 0.023

5. Secondary Outcome: Trough FVC Response at Week 4
Description: The change from baseline in Trough FVC after 4 weeks of treatment
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | -0.037 (0.033) | 0.154 (0.032) | 0.154 (0.033) | 0.150 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.191, 95% CI [0.107 to 0.275], Standard Error of Mean 0.043
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.191, 95% CI [0.106 to 0.276], Standard Error of Mean 0.043
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.187, 95% CI [0.103 to 0.270], Standard Error of Mean 0.042

6. Secondary Outcome: FVC AUC(0-3) Response
Description: The change from baseline in FVC AUC(0-3) response after 4 weeks of treatment. FVC AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in liters.
  Due to normalization the unit is liters.
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | 0.004 (0.036) | 0.257 (0.035) | 0.254 (0.036) | 0.237 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.253, 95% CI [0.160 to 0.345], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.250, 95% CI [0.156 to 0.343], Standard Error of Mean 0.047
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.233, 95% CI [0.141 to 0.325], Standard Error of Mean 0.047

7. Secondary Outcome: FVC Peak(0-3) Response
Description: The change from baseline in FVC peak(0-3) response after 4 weeks of treatment.
Time Frame: baseline and after 4 weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
Liter | 0.109 (0.038) | 0.362 (0.037) | 0.351 (0.038) | 0.335 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Olodaterol 2mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.253, 95% CI [0.155 to 0.351], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Olodaterol 5mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.242, 95% CI [0.142 to 0.341], Standard Error of Mean 0.050
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Olodaterol 10mcg - Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean for the difference = 0.226, 95% CI [0.129 to 0.324], Standard Error of Mean 0.050

8. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 0-6h (AUC 0-6h) Response After 4 Weeks
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect.
  FEV1 AUC 0-6h was calculated from 0-6 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in liters.
Time Frame: baseline and after 4weeks treatment
Population: The full analysis set (FAS) for 4 weeks treatment period which is however restricted to patients with evaluable data for this endpoint - analysis with imputation
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 78 | 80 | 79 | 85
Liter | -0.022 (0.028) | 0.090 (0.027) | 0.195 (0.027) | 0.195 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p = 0.0045, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.111, 95% CI [0.035 to 0.188], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.216, 95% CI [0.140 to 0.293], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.217, 95% CI [0.142 to 0.292], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

9. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 6-12 h (AUC 6-12h) Response After 4 Weeks
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect.
  FEV1 AUC 6-12h was calculated from 6-12 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in liters.
Time Frame: Baseline and after 4weeks treatment
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 78 | 80 | 79 | 85
Liter | -0.005 (0.028) | 0.078 (0.027) | 0.171 (0.027) | 0.186 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p = 0.0348, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI [0.006 to 0.159], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.100 to 0.252], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.190, 95% CI [0.115 to 0.265], Standard Error of Mean 0.038 — Olo 10 mcg qd minus Placebo

10. Secondary Outcome: Weekly Mean Pre-dose Morning Peak Expiratory Flow Rate (PEFR) After 4 Weeks
Description: PEFR measurements were recorded by means of a patient diary on a daily basis. This diary was used to record the twice daily PEFs,
  Morning measurements were performed immediately upon arising before administration of trial and/or rescue medication.The highest of three readings for each measurement were recorded.
Time Frame: Week 4
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 78 | 83 | 78 | 86
Liter/minute | 217.54 (4.059) | 244.80 (3.933) | 246.93 (4.059) | 254.22 (3.869)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 27.256, 95% CI [16.477 to 38.036], Standard Error of Mean 5.476 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 29.383, 95% CI [18.410 to 40.357], Standard Error of Mean 5.574 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 36.678, 95% CI [25.987 to 47.369], Standard Error of Mean 5.431 — Olo 10 mcg qd minus Placebo

11. Secondary Outcome: Weekly Mean Evening PEFR After 4 Weeks
Description: PEFR measurements were recorded by means of a patient diary on a daily basis. This diary was used to record the twice daily PEFs,
  Evening measurements were performed at bedtime.The highest of three readings for each measurement were recorded.
Time Frame: Week 4
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 78 | 83 | 78 | 86
Liter/minute | 227.39 (4.085) | 256.44 (3.955) | 258.34 (4.083) | 264.58 (3.890)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 29.052, 95% CI [18.159 to 39.946], Standard Error of Mean 5.534 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 30.955, 95% CI [19.861 to 42.049], Standard Error of Mean 5.635 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 37.191, 95% CI [26.386 to 47.996], Standard Error of Mean 5.489 — Olo 10 mcg qd minus Placebo

12. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy After 4 Weeks
Description: Weekly mean number of occasions of rescue therapy used per day (PRN salbutamol )
Time Frame: Week 4
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 83 | 79 | 86
Number of puffs | 0.778 (0.110) | 0.587 (0.107) | 0.324 (0.109) | 0.392 (0.105)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol 2mcg; Test type: Superiority or Other; p = 0.2016, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.191, 95% CI [-0.485 to 0.103], Standard Error of Mean 0.149 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol 5mcg; Test type: Superiority or Other; p = 0.0029, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.454, 95% CI [-0.752 to -0.156], Standard Error of Mean 0.151 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol 10mcg; Test type: Superiority or Other; p = 0.0095, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.387, 95% CI [-0.678 to -0.095], Standard Error of Mean 0.148 — Olo 10 mcg qd minus Placebo

13. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis, ECG and Physical Examination
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis, ECG and Physical examination. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 4 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
percentage of participants
  Atrioventricular block second degree | 0.0 | 0.0 | 0.0 | 1.2
  Blood lactate dehydrogenase increased | 0.0 | 0.0 | 1.3 | 0.0
  Blood glucose increased | 0.0 | 0.0 | 0.0 | 1.2
  White blood cell count decreased | 0.0 | 0.0 | 0.0 | 1.2

14. Secondary Outcome: Difference From Baseline in Potassium
Description: Difference from baseline in Potassium (normalized values). Normalization means that the values from different laboratories are transformed in such a way that they are directly comparable.
Time Frame: Baseline, Week 4
Population: Treated set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 79 | 84 | 79 | 86
mmol/L | 0.0 (0.5) | 0.1 (0.6) | -0.0 (0.5) | 0.1 (1.1)

15. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: Cmax only calculated if >1/3 of the patients have available pharmacokinetic parameters,thus not applicable for the Olodaterol 2 mcg
Time Frame: after first inhalated administration
Population: Treated set which is however restricted to patients with evaluable data for this endpoint (Patients in which all plasma concentration values were below limit of quantification (BLQ), were excluded from the analysis and were not included into the total number of participants affected for this outcome measure)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 53 | 81
pg/mL | 4.17 (46.7) | 8.22 (58.3)

16. Secondary Outcome: Cmax,ss (Maximum Measured Concentration of the Analyte in Plasma at Steady State)
Description: Cmax,ss only calculated if >1/3 of the patients have available pharmacokinetic parameters, thus not applicable for the Olodaterol 2 mcg
Time Frame: visit at week 4
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 67 | 78
pg/mL | 5.92 (57.4) | 13.1 (58.6)

17. Secondary Outcome: AUC0-1
Description: Area under the concentration curve from 0 to 1 hour using trapezoid rule, only calculated if >1/3 of the patients have available pharmacokinetic parameters,thus not applicable for Olodaterol 2mcg group
Time Frame: after first inhalated administration
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 30 | 77
pg*h/mL | 3.67 (35.6) | 6.08 (50.8)

18. Secondary Outcome: AUC0-1,ss
Description: Area under the concentration curve from 0 to 1 hour at steady state using trapezoid rule, only calculated if >1/3 of the patients have available pharmacokinetic parameters, thus not applicable for Olodaterol 2mcg group
Time Frame: visit at week 4
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Olodaterol 5mcg | Olodaterol 10mcg
Number analyzed (Participants) | 64 | 77
pg*h/mL | 4.85 (54.6) | 10.8 (54.0)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | Olodaterol 2mcg | Olodaterol 5mcg | Olodaterol 10mcg
Serious Adverse Events (participants affected / at risk) | 2/79 | 3/84 | 1/79 | 3/86
Other Adverse Events (participants affected / at risk) | 7/79 | 9/84 | 3/79 | 5/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Olodaterol 2mcg (N=84) | Olodaterol 5mcg (N=79) | Olodaterol 10mcg (N=86)
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Olodaterol 2mcg (N=84) | Olodaterol 5mcg (N=79) | Olodaterol 10mcg (N=86)
Nasopharyngitis (Infections and infestations) | 3 | 9 | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes